CLINICAL TRIAL: NCT07135921
Title: The Effect of Sleep Hygiene Education on Disease Management and Sleep Quality in Individuals With Cardiovascular Diseases: A Randomized Controlled Clinical Trial Protocol
Brief Title: Sleep Hygiene Education in Individuals With Cardiovascular Disease: Effects on Sleep Quality and Disease Management
Acronym: SLEEP-CARD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Deniz Talaz, Dr. Deniz Talaz, PhD, Principal Investigator, Department of Medical Nursing, Near East University, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YDU-KARD-UYKU-2025-RCT; Near East University (Other: Near East Universıty)
Record Dates: First submitted 2025-07-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Disease and Sleep Hygiene
MeSH Terms: conditions — Cardiovascular Diseases; Sleep Hygiene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Sleep Hygiene Education
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Sleep Hygiene Education — This intervention consists of a nurse-led sleep hygiene education program delivered through a 30-minute PowerPoint presentation. Participants in the intervention group will also receive twice-daily reminder messages via WhatsApp for four weeks to reinforce healthy sleep habits. The program aims to improve sleep quality and disease management in individuals with cardiovascular disease. After the study, the educational materials will also be shared with the control group.
  Arms: Intervention Group

SUMMARY:
This clinical trial aims to find out if sleep hygiene education helps people with cardiovascular disease manage their illness better and improve their sleep quality.

Participants will be randomly assigned to two groups. One group will receive sleep hygiene education through a 30-minute presentation and twice-daily reminder messages for four weeks. The other group will receive usual care without education.

Before and after the four-week period, all participants will complete questionnaires about their sleep habits, sleep quality, and disease management.

The study hopes to show that sleep hygiene education can improve participants' sleep and help them manage their disease symptoms better, leading to a better quality of life.

The trial will take place at Near East University Hospital's Cardiology Department from June to December 2025.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical diagnosis of cardiovascular disease at least one year prior
* No visual, hearing, communication, cognitive, or physical impairments
* Literate and able to use a smartphone and/or computer
* Willing to participate in the sleep hygiene education program
* Able to provide informed consent

Exclusion Criteria:

* Pregnancy
* Working night shifts
* Cognitive impairment preventing questionnaire completion
* Visual, hearing, communication, or physical impairments that prevent participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-11 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in Sleep Quality | 5 weeks (4 weeks intervention + final assessment in week 5)
  This outcome measures the change in participants' sleep quality after the 4-week sleep hygiene education program. Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI total score ranges from 0 to 21, where higher scores indicate worse sleep quality and lower scores indicate better sleep quality. Data will be collected at baseline and after completion of the intervention.

SECONDARY OUTCOMES:
Improvement in Disease Management | 5 weeks (4 weeks intervention + final assessment in week 5)
  This outcome measures the change in participants' disease self-management ability after the 4-week sleep hygiene education program. Disease management will be assessed using the Chronic Disease Self-Management Scale (CDSMS). The CDSMS total score ranges from 0 to 100, with higher scores indicating better self-management and lower scores indicating poorer self-management. Data will be collected at baseline and after completion of the intervention.